CLINICAL TRIAL: NCT03427905
Title: Autologous Adipose-Derived Adult Stromal Vascular Cell Transplantation for Alopecia
Acronym: A-ADSVC-CT-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese University (Other)
Collaborators: Reviva Regenerative Medicine Center MEIH Hospital - REVIVA PHARMACEUTICALS (for the first group) (Unknown)
Responsible Party: Principal Investigator, Nehman Makdissy, Principal Investigator, Lebanese University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTP-008-13-Ed-001
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hair Loss/Baldness; Alopecia
MeSH Terms: conditions — Alopecia | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (Active Comparator): lipoaspiration and transplantation of ADSVCs (for adipose-derived stromal vascular cells/primary fresh cells without culture) Interventions: - Procedure: Lipoaspiration; - Procedure: Transplantation
  Interventions: Procedure: Lipoaspiration
- GROUP II (Active Comparator): lipoaspiration and transplantation of ADSCs (for adipose-derived mesynchymal stem cells/after culture) Interventions: - Procedure: Lipoaspiration; - Procedure: Transplantation
  Interventions: Procedure: Transplantation

INTERVENTIONS:
Procedure: Lipoaspiration — Procedure: Lipoaspiration of fat and processing for the isolation of SVF Procedure: Transplantation
  Arms: GROUP I
Procedure: Transplantation — Procedure: Lipoaspiration of fat and processing for the isolation of SVF and culture for the obtention of ADSCS Procedure: Transplantation
  Arms: GROUP II

SUMMARY:
Most common forms of hair loss (alopecia) are caused by aberrant hair follicle cycling and changes in hair follicle morphology. However, current treatments for alopecia do not specifically target these processes. Adipose-derived stromal vascular cells (ADSVCs) that can be harvested from fat cells are one of the latest breakthroughs in the aesthetic field. The potential use of stem cell-based therapies for the repair and regeneration of various tissues and organs offers a paradigm shift that may provide alternative therapeutic solutions. This study aimed at the presentation of clinical cases to suggest a therapeutic plan comprised of acquisition of small volume of fat, followed by injection of ADSVCs in the scalp. 20 patients will be recruited for this study (considering the second group). Hair regeneration will be assessed by the pull test, hair quality, and hair density. All patients must show increased significant improvement of the hair quality and density. The obtained results must prove the efficacy and the safety of the treatment and satisfaction of the patient that will confirm the quality of the results.

DETAILED DESCRIPTION:
Hair loss is one of the most common complaints among all patients consulting a dermatologist and is usually associated with severe psychological disturbances, distress, and symptoms of depression. Most common forms of hair loss (alopecia) are caused by aberrant hair follicle cycling and changes in hair follicle morphology. Cells with stem cell properties have recently been described in many integument appendages including feathers and teeth, but the hair follicle stands out as one of the best model systems for studying adult stem cells. Hair follicles are accessible, well defined in terms of their developmental biology, and their stem cell populations are located in discrete compartments or niches.

There are three phases of hair growth, which every hair follicle undergoes. The first phase is when follicles undergo extremely rapid epithelial cell division and execute exquisitely timed differentiation programs when in the growing (Anagen) phase. The second phase is when follicles growth stops during a certain period, the (Catagen) phase. The third phase is when most follicles regress into structures that resemble immature developing follicles, after which they go into a period of mitotic quiescence, the (Telogen) phase. Stem cells are at the core of all hair dynamic events that includes a new burst of activity and further morphogenetic remodeling as the follicle grows again at the start of a new Anagen phase.

The term "Stem Cell" is given to a cell which has the ability to self-renew as well as to differentiate into defined cellular subtypes. Multipotent stem cells are present in different adult tissues such as bone marrow, dental pulp, adipose tissue, etc. and within the adipose tissue the adipose-derived stromal vascular cells (ADSVCs), which are one of the most promising stem cell population identified since the human adipose tissue is easily obtained in large quantities with little patient discomfort and secretory factors from ADSVCs have been considered as a promising therapy for skin aging. Therefore, the use of autologous ADSVCs can be promising for hair loss. Since the stromal vascular fraction (SVF) is saturated with stem cells among other cells derived from adipose tissue, cells can be called ADSVFC if they are used freshly, or ADSC/ADASC or others terms in cases of primary cells placed in culture having then the adherent feature, resulting in a set of mesenchymal stem cells (MSCs). In fact, contrary to cultured ADSCs, freshly isolated ADSVCs were shown to be highly positive for CD34, and positive for CD117 and HLA-DR. MSCs derived from adipose tissue when obtained by culture are mostly negative for CD34, and HLA-DR. This indicates clearly that primary cells are significantly more promising in cases of need to maintain a certain level of CD34 in the graft.

In the present study, the investigators aimed to use autologous ADSVCs graft for the treatment of alopecia and to assess the safety and effectiveness of the transplantation. This ADSVCs group will be compared to a group of cultured ADSCs. In fact, the study is divided into 2 groups: ADCVCs and ADSCs, where the first group had been started in 2013 and since 2016, the investigators aimed to add a comparative group by using the cultured ADSCs instead of the primary non-cultured ADSVCs. (Note: the investigators started using grafts of PRP (Platelets Rich Plasma) in 2013 before using isolated adipose-derived cells, where no significant improvement in the hair quality was observed. Then, the investigators aimed to use adipose-derived cells firstly without culture and secondly subjected to culture. The first group was done in collaboration with Reviva Regenerative Medicine Center at the Middle East Institute of Health University Hospital at Bsalim Lebanon. The second group will be realized with a collaborator to be defined by the Lebanese University after approval of the administration and corresponding committee.

The process flow is defined as following: (1) the file study: which start by receiving the file of the patient, the file will be forwarded to appointed physician coordinator for review and submission of medical report (Here Dr. Rami Anderi), then the medical report will be evaluated by the cell therapy committee and the patient will be asked for clinical examination, and after consultation a reply to the patient with medical decision will follow with an approval or not be recruited and if yes, a brief report about the procedure will be submitted and explained in details to the patient, a consent form must be signed if the patient agrees to be included in the study, (2) the patient admission: which may start by completion of the procedure forms and doing the pre-op evaluation (initial work up defined as a clinical and biological assessment upon C.A.S), followed by lipoaspiration of the subcutaneous adipose tissue to be performed by the plastic surgeon, then sample processing for isolation and characterization of the stromal vascular fraction enriched with ADSVCs (the quality control assessment will be realized before and after all the steps of the procedure starting from the SVF collection to transplantation; (3) the delivery (transplantation). The patient will be put on antibiotic/anti-inflammatory for a defined period and followed by the team at 1 week, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Hair loss
* baldness
* alopecia
* Age: ≥ 18 years
* Gender: any
* Willing to collaborate and to attend to the clinical follow-ups for four years
* Patients willing to sign informed consent
* Able and willing to comply with all study requirements
* Patients with no hereditary diseases of the hair, with no burns
* Medically suitable to undergo cell's graft surgery with local anesthesia
* Normal serum chemistry and hematology screening tests
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) serology
* No history of malignancy
* Complete history & physical examination
* Negative chest roentgenogram (CXR)
* Negative urinalysis (U/A)
* Normal thyroid exam

Exclusion Criteria:

* Patients not willing to sign informed consent
* Defects in hair scalp with a potential to affect the graft outcome
* Severe hair loss and baldness
* Infection
* Known allergy
* Known coagulation abnormalities
* Any medical condition likely interferes to cause serious adverse events during the study
* History of malignancy
* History of cognitive impairments or dementia which may impact the patient's ability to participate in the informed consent process and to appropriately complete evaluations
* Any immunodeficiency
* Any current immunosuppressive therapy other than intermittent or low dose corticosteroids
* Renal insufficiency, as defined by creatine level >1.3 mg/dL.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV
* If female, pregnancy or lactation.
* Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety or interferes with the interpretation of the study results.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of Hair loss | 6 months postoperative
  Decrease in the hair loss

SECONDARY OUTCOMES:
Improvement of hair density | 6 months postoperative
  Increase in the hair density (Trichometry) from values < 175 hair/ cm² to normal range (175 to 300 hair/ cm²)
Improvement of hair diameter | 6 months postoperative
  Increase in the hair diameter from fine hair (≤ 60 microns) to medium hair (60 to 80 microns) and thick hair (≥ 80 microns)
Improvement of the pull test | 6 months postoperative
  Decrease in the pull test measures (from 3-8 to 0-1; the number of extracted pulled hairs must be between 0 and 1 in normal patients)

CONTACTS AND LOCATIONS:
Overall Officials: Nehman Makdissy, PhD, Principal Investigator — Lebanese University; Rami Anderi, MD, Study Director — Lebanese University
Locations (1):
- Lebanese University, faculty of Sciences, section II and III, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided